CLINICAL TRIAL: NCT00434252
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Bevacizumab in Combination With Carboplatin and Paclitaxel Chemotherapy for the First-Line Treatment of Patients With Metastatic Melanoma
Brief Title: A Study of Bevacizumab With Carboplatin and Paclitaxel Chemotherapy for the First-Line Treatment of Patients With Metastatic Melanoma
Acronym: BEAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF4096g
Record Dates: First submitted 2007-02-11; First posted 2007-02-13 (Estimated); Results first posted 2011-09-28 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Melanoma
Keywords: Avastin; BEAM; Metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Carboplatin+Paclitaxel+Placebo (Placebo Comparator)
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: placebo
- Carboplatin+Paclitaxel+Bevacizumab (Experimental)
  Interventions: Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: bevacizumab — 15 mg/kg by intravenous (IV) infusion on the first day of each 3-week cycle (dose was based on patient's weight at screening and remained the same throughout study)
  Arms: Carboplatin+Paclitaxel+Bevacizumab
Drug: carboplatin — Dose based on patients' creatinine clearance (Calvert formula) and administered by intravenous (IV) infusion on the first day of each 3-week cycle, for a maximum of 10 cycles
Drug: paclitaxel — 175 mg/m^2 by IV infusion on the first day of each 3-week cycle (dose was based on patient's weight and could be adjusted for weight change)
Drug: placebo — Administered by IV infusion on the first day of each 3-week cycle
  Arms: Carboplatin+Paclitaxel+Placebo

SUMMARY:
This Phase II, multicenter, randomized, double-blind, placebo-controlled trial was designed to estimate the efficacy and characterize the safety of bevacizumab when combined with carboplatin + paclitaxel chemotherapy compared with carboplatin + paclitaxel chemotherapy alone in patients with previously untreated metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥ 18 years
* Metastatic melanoma (Stage IV)
* Histologically confirmed malignant melanoma with measurable or non-measurable disease
* Ability and willingness to comply with study and follow-up procedures

Exclusion Criteria:

* Prior treatment for Stage IV disease with chemotherapy or biologic therapy such as interferon and interleukin-2
* Complete surgical resection or irradiation of all identifiable sites of disease at randomization
* Radiation therapy within 14 days prior to Day 1
* Prior therapy with bevacizumab, sorafenib, sunitinib, or other vascular endothelial growth factor (VEGF) pathway-targeted therapy
* Melanoma of ocular origin
* Known central nervous system (CNS) disease/brain metastases (history of brain disease or active disease)
* Life expectancy of < 12 weeks
* Current, recent, or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Inadequate organ function
* History of other malignancies within 5 years of Day 1, except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications
* Inadequately controlled hypertension
* History of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Class II or greater CHF
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to Day 1
* History of hemoptysis within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Known hypersensitivity to any component of bevacizumab
* Pregnancy (positive pregnancy test) or lactation
* Current, ongoing treatment with full-dose warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schwartz, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin+Paclitaxel+Placebo: Administered by intravenous (IV) infusion every 3 weeks until disease progression, unacceptable toxicity, or for a maximum of 102 weeks, whichever occurred first. Carboplatin administration was stopped after completion of 10 treatment cycles, while paclitaxel continued to be administered with placebo.
- Carboplatin+Paclitaxel+Bevacizumab: Administered by IV infusion every 3 weeks until disease progression, unacceptable toxicity, or for a maximum of 102 weeks, whichever occurred first. Carboplatin administration was stopped after completion of 10 treatment cycles, while paclitaxel continued to be administered with bevacizumab.
Period: Overall Study
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Started | 71 | 143
Treated | 69 (One patient died and one patient withdrew prior to receiving study treatment) | 143
Completed | 7 (Continuing study drug treatment at the time of the data cutoff.) | 12 (Continuing study drug treatment at the time of the data cutoff.)
Not Completed | 64 | 131
Not completed — Lack of Efficacy | 50 | 100
Not completed — Adverse Event | 6 | 13
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 4 | 8
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab | Total
Number analyzed (Participants) | 71 | 143 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (12.6) | 59.1 (11.3) | 58.9 (11.7)
Age, Customized [Number; unit: participants]
  <= 65 years | 46 | 104 | 150
  > 65 years | 25 | 39 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 45 | 66
  Male | 50 | 98 | 148

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from randomization to documented disease progression (at least a 20% increase in the sum of the longest diameter of target lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions) or death on study (death from any cause occurring no later than 30 days after last dose of any study treatment), whichever occurred first, as determined by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST). Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From randomization up to102 weeks. As of the clinical cut-off date (April 2009), the maximum time on treatment was 88 weeks, median time was 12.4 weeks for the Placebo arm and 16.1 weeks for the bevacizumab arm.
Population: Intent-to-treat (randomized) population. For patients without documentation of disease progression or death on study, PFS was censored at the time of the last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Number analyzed (Participants) | 71 | 143
months | 4.2 [2.83 to 5.36] | 5.6 [4.21 to 6.80]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to death from any cause. Median OS was estimated using the Kaplan-Meier method. For patients without documentation of death, overall survival will be censored at the time of the last known contact.
Time Frame: Up to 102 weeks
Population: Intent-to-treat (randomized) population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Number analyzed (Participants) | 71 | 143
months | 8.6 [7.66 to 11.83] | 12.3 [10.35 to NA] — Upper limit of confidence interval not estimable due to very small number of deaths occurring after median was reached.

3. Secondary Outcome: Number of Participants With Objective Response
Description: Objective response was assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) criteria and was inclusive of complete and partial response determined on two consecutive investigator assessments conducted ≥ 4 weeks apart.
Time Frame: Up to 102 weeks
Population: Intent-to-treat (randomized) population.
Measure: Number; unit: participants
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Number analyzed (Participants) | 67 | 141
participants | 11 [7.5 to 25.3] | 36 [18.3 to 32.7]

4. Secondary Outcome: Percentage of Participants With an Objective Response
Description: Objective response was defined as a complete or partial response according to RECIST criteria as assessed by the investigator on two consecutive assessments conducted at least 4 weeks apart.
  The 95% Confidence Interval (CI) was calculated using the normal approximation to the binomial distribution.
Time Frame: Up to 102 weeks
Population: Randomized Patients with Measurable Disease at Baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Number analyzed (Participants) | 67 | 141
percentage of participants | 16.4 [7.5 to 25.3] | 25.5 [18.3 to 32.7]

5. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response was defined as the time from the initial objective response to documented disease progression or death, whichever occurred first, assessed by the investigator using RECIST. Progressive disease was defined as at least 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started, or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Duration of response was estimated using the Kaplan-Meier method.
Time Frame: Up to 102 weeks
Population: Intent-to-treat (randomized) population. Only patients with measurable disease who achieved a response (either partial or complete) were included in the analysis of duration of response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Number analyzed (Participants) | 11 | 36
months | 7.7 [3.94 to 11.56] | 6.9 [4.86 to 8.90]

6. Secondary Outcome: Six-month Landmark Survival Rate
Description: Six-month Landmark Survival Rate was defined as the percentage of participants surviving at 6 months following randomization. Overall Survival was estimated using the Kaplan-Meier method.
Time Frame: 6 months
Population: Intent-to-treat (randomized) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Number analyzed (Participants) | 71 | 143
percentage of participants | 74.6 [64.5 to 84.8] | 78.2 [71.4 to 85.0]
Statistical Analysis 1: Comparison: Carboplatin+Paclitaxel+Placebo vs Carboplatin+Paclitaxel+Bevacizumab; Test type: Superiority or Other; p = 0.5724, z-test; z-test using the standard errors computed using Greenwood's method; Difference in survival rates = 3.5, 95% CI [-8.7 to 15.7]

7. Secondary Outcome: Twenty-Four Week Landmark Stable Disease
Description: As assessed by the investigator using RECIST and defined as the absence of disease progression for 24 weeks from the time of randomization.
  The percentage of patients who did not experience disease progression or death at 24 weeks following randomization was estimated using Kaplan-Meier methodology. If no tumor assessments were performed after the baseline visit, the patient will be censored at the date of randomization plus 1 day.
Time Frame: 24 weeks
Population: Intent-to-treat (randomized) patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Number analyzed (Participants) | 71 | 143
percentage of participants | 38.0 [26.4 to 49.6] | 50.2 [41.6 to 58.7]
Statistical Analysis 1: Comparison: Carboplatin+Paclitaxel+Placebo vs Carboplatin+Paclitaxel+Bevacizumab; Test type: Superiority or Other; p = 0.0982, z-test; z-test using the standard errors computed using Greenwood's method; Difference in event rates = 12.2, 95% CI [-2.3 to 26.6]

8. Secondary Outcome: Number of Participants With Select Adverse Events
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0. Select adverse events included arterial thromboembolic events (any grade), bleeding other than pulmonary or central nervous system (CNS) bleeding (Grade >= 3), CNS bleeding (any grade), febrile neutropenia (any grade), hypertension (Grade >= 3), neutropenia (Grade >= 3), pulmonary bleeding (any grade) and wound dehiscence (Grade >= 3).
  *All serious adverse events are listed in the Adverse Event Reporting section.
Time Frame: Participants were monitored for AEs from initiation of treatment to 30 days after treatment termination.
Population: The Safety-evaluable population consisted of all patients who received at least one full or partial dose of any component of study treatment.
Measure: Number; unit: participants
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Number analyzed (Participants) | 69 | 143
participants
  Arterial thromboembolic events (any grade) | 1 | 4
  Bleeding other than pulmonary or CNS (Grade >=3) | 4 | 0
  CNS bleeding (any grade) | 0 | 1
  Febrile neutropenia (any grade) | 1 | 7
  Hypertension (Grade >= 3) | 0 | 5
  Neutropenia (Grade >= 3) | 13 | 34
  Pulmonary bleeding (any grade) | 1 | 2
  Wound dehiscence (Grade >= 3) | 0 | 2

ADVERSE EVENTS:
Time Frame: Participants were monitored for AEs from initiation of treatment to 30 days after treatment termination
Description: Safety-evaluable population. 71 patients were randomized to the Carboplatin + Paclitaxel + Placebo arm but only 69 went on to receive study treatment
  Note: The incidence of each AE/SAE is reported as the number of patients experiencing the event, not the number of occurrences for each AE/SAE.
Arm/Group | Carboplatin+Paclitaxel+Placebo | Carboplatin+Paclitaxel+Bevacizumab
Serious Adverse Events (participants affected / at risk) | 20/69 | 40/143
Other Adverse Events (participants affected / at risk) | 69/69 | 141/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin+Paclitaxel+Placebo (N=69) | Carboplatin+Paclitaxel+Bevacizumab (N=143)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 6
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Large Intestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Small Intestinal Hemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Infusion Related Reaction (General disorders) | 1 | 0
Edema Peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Sudden Death (General disorders) | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Infected Sebaceous Cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 1 | 1
Wound Infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar Hemorrhage (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Embolic Stroke (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin+Paclitaxel+Placebo (N=69) | Carboplatin+Paclitaxel+Bevacizumab (N=143)
Anaemia (Blood and lymphatic system disorders) | 17 | 23
Leukopenia (Blood and lymphatic system disorders) | 8 | 17
Neutropenia (Blood and lymphatic system disorders) | 15 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 19
Vision Blurred (Eye disorders) | 3 | 9
Visual Impairment (Eye disorders) | 4 | 5
Abdominal Pain (Gastrointestinal disorders) | 5 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 8
Constipation (Gastrointestinal disorders) | 18 | 57
Diarrhoea (Gastrointestinal disorders) | 23 | 43
Dry Mouth (Gastrointestinal disorders) | 4 | 7
Dyspepsia (Gastrointestinal disorders) | 4 | 13
Nausea (Gastrointestinal disorders) | 33 | 73
Stomatitis (Gastrointestinal disorders) | 2 | 8
Vomiting (Gastrointestinal disorders) | 18 | 33
Chills (General disorders) | 4 | 10
Fatigue (General disorders) | 51 | 102
Mucosal Inflammation (General disorders) | 0 | 11
Oedema Peripheral (General disorders) | 8 | 7
Pain (General disorders) | 7 | 18
Hypersensitivity (Immune system disorders) | 4 | 7
Sinusitis (Infections and infestations) | 1 | 10
Weight Decreased (Investigations) | 1 | 11
Anorexia (Metabolism and nutrition disorders) | 21 | 35
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 8
Dehydration (Metabolism and nutrition disorders) | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 36
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 20
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 30
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9 | 11
Dizziness (Nervous system disorders) | 6 | 20
Dysgeusia (Nervous system disorders) | 10 | 16
Headache (Nervous system disorders) | 8 | 31
Neuropathy Peripheral (Nervous system disorders) | 22 | 51
Paraesthesia (Nervous system disorders) | 5 | 11
Peripheral Sensory Neuropathy (Nervous system disorders) | 8 | 19
Anxiety (Psychiatric disorders) | 4 | 9
Depression (Psychiatric disorders) | 4 | 10
Insomnia (Psychiatric disorders) | 5 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 24
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 28
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 57
Alopecia (Skin and subcutaneous tissue disorders) | 42 | 84
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 12
Rash (Skin and subcutaneous tissue disorders) | 14 | 16
Flushing (Vascular disorders) | 2 | 11
Hypertension (Vascular disorders) | 10 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.